CLINICAL TRIAL: NCT06299007
Title: Awareness of the Need for the Evaluation of Iron Status Among Hospitalized Patients With Acute Upper Gastrointestinal Bleeding.
Brief Title: Awareness of Iron Status Evaluation in UGIB
Acronym: AISE
Status: Completed | Type: Observational
Sponsor: Hat Yai Medical Education Center (Other)
Responsible Party: Principal Investigator, Arunchai Chang, Hatyai Hospital, Hat Yai Medical Education Center
Other Study IDs: HYH EC 052-66-01; HYH EC 052-66-01 (Other Grant/Funding Number: Hatyai Hospital Education Center)
Record Dates: First submitted 2024-02-28; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: upper gastrointestinal bleeding; Anemia; iron status; iron deficiency
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Anemia; Iron Deficiencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients who were admitted due to upper gastrointestinal bleeding and had anemia

SUMMARY:
BACKGROUND: Data on the awareness of the need to evaluate iron status and IDA prevalence in acute UGIB are limited.

OBJECTIVES: This study aimed to investigate the rate of evaluation of iron status and prevalence of iron deficiency anemia (IDA) and the associated factors in patients with anemia hospitalized for acute upper gastrointestinal bleeding (UGIB).

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years of age who were admitted because of acute UGIB and were diagnosed with anemia from UGIB during hospitalization.

Exclusion Criteria:

* patients who had previously undergone endoscopy at another institution before admission
* patients who had a definite cause of UGIB that was inconclusive
* incomplete data for analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who were admitted because of acute UGIB at Hatyai Hospital between January 2016 and December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 867 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
iron status measurement | During admission
  iron status measurement during admission among patients hospitalized for acute UGIB.

SECONDARY OUTCOMES:
Iron deficiency anemia | During admission
  patients with anemia who had serum ferritin < 30 μg/L and/or transferrin saturation < 16%.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatyai Hospital, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barkun AN, Almadi M, Kuipers EJ, Laine L, Sung J, Tse F, Leontiadis GI, Abraham NS, Calvet X, Chan FKL, Douketis J, Enns R, Gralnek IM, Jairath V, Jensen D, Lau J, Lip GYH, Loffroy R, Maluf-Filho F, Meltzer AC, Reddy N, Saltzman JR, Marshall JK, Bardou M. Management of Nonvariceal Upper Gastrointestinal Bleeding: Guideline Recommendations From the International Consensus Group. Ann Intern Med. 2019 Dec 3;171(11):805-822. doi: 10.7326/M19-1795. Epub 2019 Oct 22. PMID 31634917
- [Background] Stein J, Connor S, Virgin G, Ong DE, Pereyra L. Anemia and iron deficiency in gastrointestinal and liver conditions. World J Gastroenterol. 2016 Sep 21;22(35):7908-25. doi: 10.3748/wjg.v22.i35.7908. PMID 27672287
- [Background] Kulnigg S, Stoinov S, Simanenkov V, Dudar LV, Karnafel W, Garcia LC, Sambuelli AM, D'Haens G, Gasche C. A novel intravenous iron formulation for treatment of anemia in inflammatory bowel disease: the ferric carboxymaltose (FERINJECT) randomized controlled trial. Am J Gastroenterol. 2008 May;103(5):1182-92. doi: 10.1111/j.1572-0241.2007.01744.x. Epub 2008 Mar 26. PMID 18371137
- [Background] Cotter J, Baldaia C, Ferreira M, Macedo G, Pedroto I. Diagnosis and treatment of iron-deficiency anemia in gastrointestinal bleeding: A systematic review. World J Gastroenterol. 2020 Dec 7;26(45):7242-7257. doi: 10.3748/wjg.v26.i45.7242. PMID 33362380